CLINICAL TRIAL: NCT02134769
Title: Incidence of Catheter-related Bloodstream Infections Using Bionecteur Device
Brief Title: Influence of Bionecteurs on Catheter-associated Infection
Acronym: Bionect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Vygon GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIONECT-2014; ZVK-Bionect (Other: University Hospital Tuebingen)
Record Dates: First submitted 2014-04-09; First posted 2014-05-09 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2015-07

CONDITIONS: Infection
Keywords: catheter-related bloodstream infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No use of Bionecteur; handling according to institutional guideline
- Bionecteur (Active Comparator): Use of Bionecteur; handling according to institutional guideline
  Interventions: Device: Bionecteur

INTERVENTIONS:
Device: Bionecteur — Using Bionecteur at each lumina of the catheter; handling according to institutional guideline
  Other Names: bionector® company: Vygon
  Arms: Bionecteur

SUMMARY:
Bionecteur® is a protective non-touch applicator to ensure aseptic connection made by Vygon. However, there are no studies describing a positive effect of using Bionecteurs ® in regard to catheter-related bloodstream infections. In this study Bionecteur® will be used on central venous lines and arterial lines in postoperative patients of a 40-bed ICU. The incidence of catheter-related bloodstream infections will we compared to patients without inclusion of Bionecteur® devices.

DETAILED DESCRIPTION:
* Prospective, randomised observational study
* Postsurgical patients in an anesthesiological ICU with ICU LOS (LOS: length of stay) > 3 days

  * Inclusion:

    ---- Age ≥ 18 years

    ---. demand of central venous and arterial line

    --- written consent of patient and/or assignee
  * Exclusion

    * Handicapped patients
    * patient with ICU LOS < 3 days
* Study design

  1. Three days after admission to ICU blood cultures are drawn to exclude preexisting blood stream infection
  2. Patients in a bed with even number are assigned to Bionecteur® group. Control group (without using bionecteurs) are patients with an odd bed number.
  3. Biconecteurs® are connected to all lumens of the central catheter and to arterial catheter. Control group is treated without using Bionecteurs®. Handling of vascular catheters are performed as described in institutional guidelines in both groups.
  4. Catheter-related bloodstream infections are monitored by an independent person during ICU treatment
  5. The study will be finished ab discharge of ICU or removal of catheters.

ELIGIBILITY:
Inclusion Criteria:

* Length of Stay (LOS) in ICU > 3 days
* written consent by patient or notarial carers
* medical indication for central venous line/arterial line

Exclusion Criteria:

* handicap
* LOS ICU < 3 days
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-related bloodstream infections using Bionecteurs | 1 year

SECONDARY OUTCOMES:
Length of Stay in ICU | 1 year
  Determine days in ICU with centrral venous catheter

CONTACTS AND LOCATIONS:
Overall Officials: Helene A Haeberle, MD, Principal Investigator — University Hospital Tuebingen, Germany
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koeppen M, Weinert F, Oehlschlaeger S, Koerner A, Rosenberger P, Haeberle HA. Needle-free connectors catheter-related bloodstream infections: a prospective randomized controlled trial. Intensive Care Med Exp. 2019 Dec 2;7(1):63. doi: 10.1186/s40635-019-0277-7. PMID 31792889